CLINICAL TRIAL: NCT05247398
Title: Mechanisms of a Dynamic Stability Approach
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OT-2021-30466; UL1TR002494 (NIH); KL2TR002492 (NIH)
Record Dates: First submitted 2022-01-27; First posted 2022-02-18 (Actual); Results first posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Thumb Carpometacarpal Osteoarthritis; Thumb Basal Joint Osteoarthritis
Keywords: Arthritis; Exercise; Thumb; Treatment; Intervention; Dynamic stability; Hand; Therapy; Occupational; Physical
MeSH Terms: conditions — Arthritis; Motor Activity

STUDY DESIGN:
Intervention Model Description: prospective pre-postinterventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dynamic Stability Exercise Program (Experimental): Involves four 60-minute occupational therapy visits as well as a daily home program across a 8-week period. Clinic visits focus primarily on home program coaching, and progression of the exercise regimen. Home programs involve daily exercises which follow the intensity and duration recommended for older adults. The intervention focuses on enhancing mobility and strength of the thumb for use during daily activities.
  Interventions: Other: Dynamic Stability Exercise Program

INTERVENTIONS:
Other: Dynamic Stability Exercise Program — The thumb CMC DS intervention involves four 60-minute occupational therapy visits as well as a daily home program across a 8-week period. Clinic visits focus primarily on home program coaching, and progression of the exercise regimen. Home programs involve daily exercises which follow the intensity and duration recommended for older adults.

SUMMARY:
Background. Arthritis is the leading cause of disability in the United States and osteoarthritis (OA) of the hand affects an estimated 25.6 US residents. OA of the thumb carpometacarpal (CMC) joint is the most disabling form of hand OA. Rehabilitation for persons with thumb CMC OA is recommended as the initial treatment and often involves instruction on joint protection and fitting of a splint to reduce joint stress and pain. More recently, evidence has suggested that specialized exercise may impact a factor linked to this condition, altered joint mechanics. Health records data also suggests that these exercises reduce pain and disability more than what would be experienced by those receiving standard care (SOC) rehabilitation. However, there has not yet been a prospective investigation on how these dynamic stability (DS) exercises alter joint mechanics, improve function, and reduce pain relative to standard treatment. Relatedly, thumb CMC mechanics are most often assessed by physicians through CAT scan and although rehabilitation therapists are not licensed to conduct such assessments, they could benefit from 'real-time' imaging to inform and evaluate the mechanical effects of treatment. Sonography might afford therapists the precision to evaluate mechanical response to treatment yet it is not yet known if thumb CMC sonography corresponds with the gold standard, CAT scan.

Goal and Specific Aims. The long term goal this line of study is to reduce the effects of thumb CMC OA on activity performance and participation through non-invasive and non- pharmacological interventions. We expect to achieve our goals by pursuit of the following two specific aims: 1). Determine if a novel exercise regimen reduces radiographic thumb CMC joint misalignment among persons with thumb carpometacarpal osteoarthritis and 2) Evaluate the accuracy of ultrasound compared with CAT scan (reference standard) for quantifying thumb CMC subluxation

Design and Methods. Specific aim 1 will be addressed through a prospective pre-post interventional study of a 8-week clinic-based dynamic stability program and will undergo a CAT scan before treatment and upon completion of the program (9 weeks) and specific aim 3 will be addressed through a psychometric 'concurrent validity' design.

ELIGIBILITY:
Inclusion Criteria:

* adults with radiographically-confirmed thumb CMC OA

Exclusion Criteria:

* Persons who have had cortisone treatments to the affected thumb within the prior three months, thumb CMC joint replacement, inflammatory arthritis, Ehlers Danlos Syndrome, Marfan's disease, pregnancy or questionable pregnancy, cognitive disorders which would preclude a client from following the testing commands and home program participation, concomitant conditions affecting the arthritic thumb, grade 4 arthritis staging, no ongoing hand rehabilitation (i.e., within prior 6 months), non-English Speaking, and pain which precludes participants from completing testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey McGee, Principal Investigator — UMN
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dynamic Stability Exercise Program
Started | 21
Completed | 20
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dynamic Stability Exercise Program
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Subluxation of Thumb Carpometacarpal Joint as Per CAT Scan
Description: CAT scan will be used at baseline and 9 weeks to obtain measurements as per the American College of Radiology's 2013 Technical Standards. A validated positioning jig reproduced by our lab will be used to maintain standardized joint positioning and standardize stress to the thumb metacarpal during fluoroscopic examination. "Joint subluxation" is a measure of thumb CMC instability and will be measured in millimeters.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Dynamic Stability Exercise Program
Number analyzed (Participants) | 20
millimeters | .66 (.99)

2. Primary Outcome: Subluxation of Thumb Carpometacarpal Joint as Per CAT Scan
Description: as for outcome 1
Time Frame: 9 weeks post intervention
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Dynamic Stability Exercise Program
Number analyzed (Participants) | 20
millimeters | .24 (.77)

3. Primary Outcome: Subluxation of Thumb Carpometacarpal Joint as Per Sonography
Description: Sonographic assessment of thumb carpometacarpal subluxation will occur at the time of participants' baseline CAT scan. The same views, position jig and standardized upper limb postures used for the fluoroscopic assessments will again be employed. The thumb CMC joint sonographic procedures described by Oo et al. and the general guidelines put forth by American Institute of Ultrasound in Medicine will be followed. Long axis views of the dorsal and radial borders of the thumb CMC joint will be visualized via use of the Philips Lumify Portable Sonography Device. In these views, the amount of translation of metacarpal base with respect to trapezium will be quantified in millimeters
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Dynamic Stability Exercise Program
Number analyzed (Participants) | 20
millimeters | .92 (1.3)

4. Secondary Outcome: Michigan Hand Questionnaire
Description: Disability was measured with the Michigan Hand Outcomes Questionnaire (MHQ), an upper extremity-specific self-report questionnaire assessing symptomology and disability across 6 domains: hand function, activities of daily living, work performance, satisfaction, aesthetics/cosmesis, and pain. Right- and left-hand total and subscale scores are produced. Scores range from 0-100, with higher total scores and scores across the first 5 subscales indicating greater abilities or better results, and lower scores on the last subscale indicating less pain. The MHQ has high reliability, validity, and responsiveness among adults with upper extremity rheumatic conditions including OA. For this study, only the total score of the affected hand was reported. Given the high prevalence of bilateral CMC1 OA, the total score from the dominant hand was selected when bilateral CMC1 OA was present.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dynamic Stability Exercise Program
Number analyzed (Participants) | 20
score on a scale | 58.9 (16.6)

5. Secondary Outcome: Michigan Hand Questionnaire
Description: Disability was measured with the Michigan Hand Outcomes Questionnaire (MHQ), an upper extremity-specific self-report questionnaire assessing symptomology and disability across 213 6 domains: hand function, activities of daily living, work performance, satisfaction, aesthetics/cosmesis, and pain. Right- and left-hand total and subscale scores are produced. Scores range from 0-100, with higher total scores and scores across the first 5 subscales indicating greater abilities or better results, and lower scores on the last subscale indicating less pain. The MHQ has high reliability, validity, and responsiveness among adults with upper extremity rheumatic conditions including OA. For this study, only the total score of the affected 219 hand was reported. Given the high prevalence of bilateral CMC1 OA, the total score from the dominant hand was selected when bilateral CMC1 OA was present.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dynamic Stability Exercise Program
Number analyzed (Participants) | 20
score on a scale | 76.5 (12.9)

6. Secondary Outcome: Numerical Pain Rating
Description: Pain severity was measured with a 0-10 Numerical Pain Rating Scale (NPRS), from which participants rated their pain intensity during daily activities over the last 24 hours, with 0 indicating no pain and 10 indicating the worst imaginable pain. The NPRS was selected because it has been established as a clinically relevant tool in persons with various rheumatic diagnoses including CMC1 OA.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dynamic Stability Exercise Program
Number analyzed (Participants) | 20
score on a scale | 4.4 (2.3)

7. Secondary Outcome: Numerical Pain Rating
Description: as for outcome 6
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dynamic Stability Exercise Program
Number analyzed (Participants) | 20
score on a scale | 2.3 (1.4)

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Dynamic Stability Exercise Program
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

LIMITATIONS AND CAVEATS:
Fluoroscopic measurements were initially planned rather than CAT but the instrumentation proved unreliable and inaccessible. CAT imaging offered a more robust and reliable solution but additional time was needed for procedural changes and IRB approval. While CAT data affords opportunities for more rigorous assessment of joint kinematics, the negligible joint space found within the thumbs of many participants has slowed our capacity to segment the images when preparing 3D models.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT05247398/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT05247398/ICF_001.pdf